CLINICAL TRIAL: NCT07252180
Title: A Prospective Study Comparing Patient Satisfaction and Efficacy of Two Different Methods of Ablation of Inlet Patches: Argon Plasma Coagulation Versus Radio Frequency Ablation
Brief Title: Comparing Two Different Methods of Ablation of Inlet Patches (APC vs RFA)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0190-25-ASF
Record Dates: First submitted 2025-11-19; First posted 2025-11-26 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: GERD (Gastroesophageal Reflux Disease); Throat Disorders
Keywords: inlet patch; GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Argon Plasma Coagulation

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into 1 of 2 treatment arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APC (Active Comparator): Argon plasma coagulation (APC) will be used to ablate the inlet patch
  Interventions: Procedure: Argon plasma coagulation (APC)
- RFA (Active Comparator): Radio frequency ablation (RFA) will be used to ablate the inlet patch
  Interventions: Procedure: RFA

INTERVENTIONS:
Procedure: Argon plasma coagulation (APC) — During upper endoscopy, the inlet patches with be ablated. One arm with undergo APC ablation while the other arm will undergo RFA ablation.
  Arms: APC
Procedure: RFA — Patients with have the inlet patch treated by RFA
  Arms: RFA

SUMMARY:
The goal of this prospective study is to compare 2 different treatment options for the ablation of inlet patches in patients with esophageal symptoms. The main questions it aims to answer are:

Is 1 method more effective than the other? Do patients prefer 1 method over the other?

Participants will undergo ablation with either argon plasma or radiofrequency.

DETAILED DESCRIPTION:
Inlet patches (IP) are areas of ectopic gastric mucosa in the proximal esophagus. [1-4] They also been referred to as cervical inlet patch (CIP), heterotopic gastric mucosa (HGM), heterotopic gastric mucosa of the proximal esophagus (HGMPE), and heterotopic gastric mucosa of the upper esophagus (HGMUE). While initially thought to be rare, they are in fact frequently found. Recent studies, including those specifically evaluating for their presence, have found IP in 10-14% of patients undergoing endoscopy [5-10].

While frequently identified as an incidental lesion, there is growing data that IP can cause symptoms, many of which are attributed to their ability to produce acid [11-13]. A recent meta-analysis comparing patients with IP to those without IP identified heartburn, dysphagia, throat discomfort, globus, hoarseness, and cough as being more prevalent in patients with IP [14].

Studies have shown that some throat symptoms have improved with ablation of IP performed during upper endoscopy [15-23]. The initial prospective studies involved treatment using argon plasma coagulation (APC) and showed safety, effective ablation of the IP, and improvement in symptoms [15-17]. Similar results have been shown in more recent larger retrospective studies [18,19], as well as in pediatric populations [20,21]. While most studies used APC to ablate IP, some studies also showed that radio frequency ablation (RFA) was successful in eradicating IP and improving symptoms [22,23]. However, to date, no studies have compared these two ablative methods.

In the investigators' experience, they have successfully used both methods to ablate IP. However, several patients have complained of sore throats after APC ablation, and the investigators have not experienced this after RFA. Additionally, in prior studies, patient satisfaction with these procedures has not been explored.

Aims The aims are to compare two proven methods of ablating IP-APC and RFA. The primary endpoint will be to compare patient satisfaction with the procedures (rated on a 0-10 scale), as well as complaints of pain or discomfort afterwards. Secondarily, the investigators will compare the efficacy of ablation between the two methods in terms of the number of sessions required to achieve complete IP eradication. Finally, the investigators will also assess differences in symptom improvement between the two groups.

Methods Study design and patients This will be a prospective, randomized, single-blinded study. Patients with known IP (at least 5 mm in size) will be included. IP diagnosis will be based on its typical endoscopic appearance. Confirmation by pathology will not be necessary. Patients will need to have symptoms suggesting that the IP is symptomatic and that ablation is indicated. Symptoms include globus sensation, sore throat, cough, hoarseness, or dysphagia. Patients will complete the Reflux Symptom Index (RSI) regarding their symptoms (see below).[24] The RSI is a validated questionnaire assessing nine different aspects of throat symptoms possibly related to acid reflux. Patients will then be randomized to receive either of the two treatment methods (APC or RFA). Patients will be blinded as to which ablation method will be performed.

Treatment methods During standard upper endoscopy, the IP will be ablated per standard protocol. For APC, this includes a power flow of 60W with argon flow set at 2 L/min. [16] The APC catheter will be inserted via the endoscope and ablations will be performed until the entire IP is ablated.

For RFA, the through-the-scope RFA device with be used with an energy density setting of 12 J/cm2.[22] The probe will be inserted via the endoscope and three deliveries of energy will be applied to the IP.

Treatment safety and literature on the subject are detailed in the investigator's brochure.

Additional study components Five days after the endoscopy, patients will be called to assess how they are feeling. This will include questions to assess their satisfaction with the procedure (0-10) and any throat pain or discomfort (0-10). Additionally, they will be asked if they required any pain medication or had any doctor's visits regarding pain/discomfort.

One month after the initial procedure, patients will return for a repeat upper endoscopy. This will be to assess whether complete eradication of the IP was achieved. If residual IP is seen, then a repeat ablation will be performed with the same method as the initial procedure. Prior to the procedure, patients will again complete the RSI to see if there has been any change in their symptoms.

If residual IP is noted on the second endoscopy, then another procedure will be repeated in another month. The investigators will perform up to 3 ablation procedures, which should result in complete ablation in most patients. (See details with literature on the subject in the investigator's brochure). Each time, symptoms will be reassessed via the RSI as previously described.

Outcomes and statistical analysis The main outcome will be the patient satisfaction score assessed five days after the initial ablation. This score (0-10) will be compared between the two groups.

Additional secondary variables that will be compared include: the percentage with pain or requiring medication after the procedure; the number of procedure sessions required to achieve complete IP eradication; and the changes in overall symptom scores (RSI) after ablation has been achieved.

Continuous variables will be compared by using t-tests or the Mann-Whitney U test (depending on the normality of the distribution). Categorical variables will be compared by using the Chi-square test or Fischer's exact test (depending on the number of results). For all statistical calculations, a p-value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Inlet patch >5 mm in size
* Esophageal or throat symptoms
* Willing to participate

Exclusion Criteria:

* No inlet patch
* Unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | 5 days after intervention
  The main outcome will be the patient satisfaction score assessed five days after the initial ablation. This score will be on a 0-10 scale where 0 represents a horrible experience and 10 represents a wonderful experience. This score will be compared between the two groups.

SECONDARY OUTCOMES:
Procedures to eradication | 1 month after interventions
  The number of procedure sessions required to achieve complete IP eradication
Improvement in symptoms | 1 month after interventions
  The changes in overall symptom score, assessed via the Reflux Symptom Index (RSI), after ablation has been achieved. The RSI contains 9 symptom domains, each of which is scored between 0 (no symptoms) and 5 (severe symptoms), for a range in total scores between 0 and a maximum of 45.

CONTACTS AND LOCATIONS:
Locations (1):
- Shamir Medical Center, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rusu R, Ishaq S, Wong T, Dunn JM. Cervical inlet patch: new insights into diagnosis and endoscopic therapy. Frontline Gastroenterol. 2018 Jul;9(3):214-220. doi: 10.1136/flgastro-2017-100855. Epub 2017 Nov 9. PMID 30046427
- [Background] Chong VH. Clinical significance of heterotopic gastric mucosal patch of the proximal esophagus. World J Gastroenterol. 2013 Jan 21;19(3):331-8. doi: 10.3748/wjg.v19.i3.331. PMID 23372354
- [Background] von Rahden BH, Stein HJ, Becker K, Liebermann-Meffert D, Siewert JR. Heterotopic gastric mucosa of the esophagus: literature-review and proposal of a clinicopathologic classification. Am J Gastroenterol. 2004 Mar;99(3):543-51. doi: 10.1111/j.1572-0241.2004.04082.x. PMID 15056100